CLINICAL TRIAL: NCT00732251
Title: An Open Label, Naturalistic Study With Allopurinol Augmentation for Prevention of Mania in Bipolar Disorder
Brief Title: Allopurinol Maintenance Study for Bipolar Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The outpatient area of the department of psychiatry at CSMC closed.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: West Coast College of Biological Psychiatry Inc (Unknown)
Responsible Party: Principal Investigator, Itai Danovitch, Chairman, Department of Psychiatry, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB13414
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Bipolar Disorder; Mania; Mixed Mania
Keywords: Bipolar Disorder; Stable Bipolar Disorder; Mania; Mixed mania; Allopurinol
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allopurinol (Experimental): Using an open label, naturalistic design, subjects will continue with their current psychiatric medications during the study. Allopurinol will be given at a fixed dose of 300 mg/day for the first week and then 600mg/d for the remainder of the study. Subjects who cannot tolerate the 600mg dose will be given a dose of 300mg/d. Subjects will participate in monthly follow up visits for 24 months. Subjects who develop a substance abuse or substance dependence disorder during the study will be terminated from the study. Also, subjects who develop a medical condition which can affect their mood stability will be terminated from the study.
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — Allopurinol: 300-600 mg/day over a 24 month period
  Other Names: Zyloprim, Aloprim

SUMMARY:
The purpose of this study is to investigate the efficacy of allopurinol as an augmentation agent for the prevention of mania in bipolar disorder patients with currently stable mood.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the efficacy of allopurinol as an augmentation agent for the prevention of mania in bipolar disorder patients with currently stable mood. Bipolar disorder is a mental disorder with severe mood swings (mania and depression). Despite the development of medications for mania, they may have significant side effects, high costs and the need for serum level monitoring. These factors adversely affect medication compliance in bipolar patients. One recent study indicated the efficacy of allopurinol in the treatment of bipolar mania. Our hypothesis is that the addition of allopurinol to standard medications for bipolar disorder will decrease the recurrences of manic episodes compared to standard medications.

This study will recruit bipolar disorder patients currently mood stable on a therapeutic dose of an anti-manic medication. Stable mood will be defined as a Young Mania Rating Scale score ≤10 and Hamilton Depression Rating Scale ≤10. Subjects must have a diagnosis of bipolar disorder confirmed by the Mini International Neuropsychiatric Interview. Young Mania Rating Scale and Mini International Neuropsychiatric Interview are common research questionnaires used in bipolar disorder studies. Potential subjects will be identified and approached during an outpatient clinical visit by a member of the research team and identified by their treating physicians and referred to the researchers.

This study involves adding allopurinol to subjects' current bipolar medications. This study will be a open label, naturalistic study. The subject will be examined monthly for manic symptoms for 2 years. Semi-structured interviews and study questionnaires will be administered to subjects at each visit. Monthly Follow-up Study Visits (once per month for 2 years - Months 1-5, 7-11, 13-17, 19-23) may be conducted either in-person or over the phone. All of the questionnaires will be administered by a clinician if the visit is completed over the phone. However, the 6-month interval visits (Months 6, 12, 18, and 24) must be done at the research center.

The primary outcome measure will be the number of manic episodes in the 2 year study period. A manic episode will be defined by a Young Mania Rating Scale score ≥20.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between ages 18 and 70.
2. Subjects must meet diagnostic and statistical manual of mental disorders 4th edition criteria for bipolar disorder confirmed by the Mini International Neuropsychiatric Interview.
3. Subjects must be taking at least one medication for mania at a therapeutic dose for at least 2 weeks.
4. Subjects must have been diagnosed with bipolar disorder, type 1, for at least 2 years prior to baseline.
5. Subjects must have adequate response to medications as evidenced by Young Mania Rating Scale score less than or equal to 10 at screening and at baseline.
6. Subjects must have adequate response to medications as evidenced by Hamilton Depression Rating Scale score less than or equal to 10 at screening and at baseline.
7. Subjects must have had at least 1 manic episode in the 2 year period prior to entering the study.
8. Female subjects must be either postmenopausal for at least 1 year, surgically sterile, abstinent or practicing an effective method of birth control if sexually active. Acceptable methods of birth control during this study are regular use of contraceptive pills, intra-uterine devices, barrier methods or abstinence. Female subjects must also have a negative urine pregnancy test at screening, baseline and other time points throughout the study.
9. Subjects must be able and willing to comply with self-administration of medication or have consistent help/support available.
10. Subjects must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
11. Subjects must be able and willing to meet or perform study requirements (e.g. answer self-administered questionnaires).
12. Subjects must be willing to allow study staff to contact subject's regular psychiatrist while the subject is in the study.

Exclusion Criteria:

1. Subjects who are unable to provide informed consent.
2. Subjects with a serious, unstable medical illness (such as cardiovascular, respiratory, neurologic, hematologic, renal, hepatic, endocrine, immunologic, or other systemic illness), a history of cerebrovascular disease, uncontrolled diabetes mellitus or acquired immunodeficiency syndrome (AIDS). Subjects with chronic illness must be stable and otherwise physically healthy on the basis of a physical examination, medical history, electrocardiogram and the results of blood biochemistry, hematology tests and a urinalysis.
3. Subjects who develop a medical condition during participation which can affect mood stability (i.e. seizure disorder, brain tumors, brain trauma, stroke, multiple sclerosis, etc.)
4. Subjects who develop substance abuse or dependence during participation in the study.
5. Subjects taking azathioprine, mercaptopurine, apalcillin, and/or amoxicillin.
6. Subjects who have been intoxicated with alcohol or drugs within the last 72hrs.
7. Subjects with a history of severe pre-existing gastrointestinal narrowing or inability to swallow oral study medication whole with the aid of water.
8. Female subjects who are pregnant or nursing.
9. Subjects who have previously participated in this study.
10. Subjects with an anticipated life expectancy of 6 months or less.
11. Subjects who have received an experimental drug or used an experimental medical device within 1 month of screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Itai Danovitch, MD, Study Chair — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- See also: Cedars-Sinai Medical Center Website — http://www.csmc.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 subjects screen failed.
Period: Overall Study
Arm/Group | Allopurinol
Started | 8
Completed | 1
Not Completed | 7
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 3
Not completed — Early Term due to Site Closure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Allopurinol
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Manic Episodes According to the Young Mania Rating Scale
Description: Young Mania Rating Scale is an 11-item, clinician-administered scale to assess severity of manic symptoms before, during and after treatment. Four items are graded on a min. 0 to max. 8 scale (irritability, speech, thought content and disruptive/aggressive behavior) while the remaining 7 items are graded on a min. 0 to max. 4 scale. A score of 0 indicates behavior is absent and score of 4 or 8 indicates the behavior is present and severe.
  The change in score between Baseline and the Completion Visit will be reported. Ideally, the two time points will be Baseline and 6 Weeks after Baseline, but if a subject terminates early, the last Young Mania Rating Scale score will be used. The scores from each question are added for a total score ranging from min. 0 to max 60; higher scores indicate greater severity of symptoms. A score of 0-12 indicates the absence of mania or a very mild manic state, a score of 13-20 or higher indicates a mild manic episode, and over 20 indicates a manic state.
Time Frame: 2 Years
Population: The outcome measure will be the total number of patient visits at which the Young Mania Rating Scale was administered per the number of patient visits at which a manic episode (according to the Young Mania Rating Scale) was recorded. The number of manic episodes prior to study start were not collected.
Measure: Count of Units; unit: patient visits
Units Other Than Participants: patient visits
Arm/Group | Allopurinol
Number analyzed (Participants) | 8
Number analyzed (patient visits) | 81
patient visits | 3

2. Secondary Outcome: Number of Depressive Episodes Per Patient Visit According to the Hamilton Depression Scale
Description: The Hamilton Depression Rating Scale is a tool used to determine a patient's level of depression before, during, and after treatment. The Hamilton Depression Scale form lists 21 items, but the scoring is based on the first 17 questions. Eight items are scored on a 5-point scale, ranging from 0 (min) = not present to 4 (max) = severe. Nine are scored from 0 (min) to 2 (max). The sum of the scores from the first 17 questions is: 0 (min) to 7 (max) = normal, 8 (min) to 13 (max) = mild depression, 14 (min) to 18 (max) = moderate depression, 19 (min) to 22 (max) = severe depression and ≥ 23=very severe depression. A score of 11 or more indicates a depressive episode in terms of this outcome measure.
Time Frame: 2 years
Population: Total number of patient visits at which the Hamilton Depression Scale was administered per the number of patient visits at which a depressive episode (according to the Hamilton Depression Scale) was recorded. The number of depressive episodes prior to the study were not collected.
Measure: Count of Units; unit: patient visits
Units Other Than Participants: patient visits
Arm/Group | Allopurinol
Number analyzed (Participants) | 8
Number analyzed (patient visits) | 86
patient visits | 7

3. Secondary Outcome: Number of Psychiatric Hospitalizations
Description: The number of psychiatric hospitalizations that occur during the study will be compared to the number of hospitalizations that occurred prior to the study.
Time Frame: 2 years
Population: Data on the number of hospitalizations was not collected before or during the study
Units Other Than Participants: hospitilizations
Arm/Group | Allopurinol
Number analyzed (Participants) | 0
Number analyzed (hospitilizations) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Allopurinol
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allopurinol (N=8)
Hospitalization (Psychiatric disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes